CLINICAL TRIAL: NCT04695418
Title: Effectiveness of Rice Germ Supplementation on Body Composition, Metabolic Parameters, Satiating Capacity and Amino Acid Profiles in Obese Postmenopausal Women: a Pilot Randomized Controlled Clinical Trial
Brief Title: Effectiveness of Rice Germ Supplementation on Body Composition, Metabolic Parameters, Satiating Capacity and Amino Acid Profiles in Obese Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1402/22052019
Record Dates: First submitted 2020-12-29; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Obesity
Keywords: Rice Germ; Body composition; Amino acids
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): an isocaloric wheat germ-based supplement
  Interventions: Combination Product: Placebo
- Rice Germ (Active Comparator)
  Interventions: Dietary Supplement: Rice Germ

INTERVENTIONS:
Dietary Supplement: Rice Germ — The rice germ was taken every day (25 g in the morning with breakfast and 25 g in the afternoon as snacks) for four weeks
  Arms: Rice Germ
Combination Product: Placebo — An isocaloric wheat germ-based supplement was taken every day (25 g in the morning with breakfast and 25 g in the afternoon as snacks) for four weeks
  Arms: Placebo

SUMMARY:
Rice germ (RG) may be a safe and effective dietary supplement for obesity in menopause, considering its high protein content and considerable amounts of essential amino acids, good fatty acids, and fiber. This pilot randomized, blinded, parallel group, placebo-controlled pilot trial investigated the effectiveness of four weeks of RG supplementation (25 g twice a day) on body composition, measured by Dual Energy X-Ray Absorptiometry (DXA), as primary outcome, and metabolic parameters, amino acid profiles and satiating capacity, as secondary outcomes, in obese postmenopausal women following a tailored hypocaloric diet (25-30% less than daily energy requirements). Twenty-seven women were randomly assigned to the supplemented group (14) or placebo group (13). There was a significant interaction between time and group for body mass index (BMI) (p<0.0001), waist (p=0.002), and hip circumference (p=0.01), total protein (0.008), albumin (0.005), Homeostasis Model Assessment index (p=0.04), glycine (p=0.002), glutamine (p=0.004), and histidine (p=0.007). Haber's means over time showed a clearly greater feeling of satiety for the supplemented compared to the placebo group. These findings indicate that RG supplementation in addition to a tailored diet counterbalanced the metabolic changes typical of menopause, with improvements in BMI, body composition, insulin resistance, amino acid profiles and satiety.

ELIGIBILITY:
Inclusion Criteria:

* obesity (BMI 30-40 kg/m2)
* age 50-65
* menopause
* sedentary women and non-smoking,
* women who did not drink more than six glasses (one glass: 125 mL) of wine a week and did not drink hard liquor (alcohol content at least 20% alcohol by volume)
* women who agreed not to take part in any other weight loss program

Exclusion Criteria:

* evidence of heart, kidney or liver disease
* women who met the Diagnostic and Statistical Manual-IV (DSM-V) criteria for a current diagnosis of major depressive disorder
* taking any medications for weight loss
* control of cholesterol and triglycerides for anti-inflammatory purposes
* pregnancy
* lactating
* Type 1 diabetes mellitus, irritable bowel disease, celiac disease, chronic pancreatitis
* antibiotic use in the last three months
* probiotic/prebiotic treatment in the last four weeks.

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-01-28 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-27 (Actual)

PRIMARY OUTCOMES:
Change of body composition | Baseline and 4 weeks
  free fat mass (g), fat mass (g), visceral abdominal tissue (g)

SECONDARY OUTCOMES:
Change of amino acid profiles | Baseline and 4 weeks
  aspartic acid, glutamic acid, alanine, arginine, asparagine, cysteine, citrulline, phenylalanine, glycine, glutamine, isoleucine, histidine, methylhistidine, methionine, ornithine, serine, tyrosine, threonine, tryptophan, valine (micromol/L)
Change of biochemical metabolic parameters | Baseline and 4 weeks
  total serum cholesterol, triacylglycerol, HDL-cholesterol, LDL-cholesterol, apolipoprotein A, apolipoprotein B, glucose, prealbumin, iron, uric acid, creatinine, electrolytes (mg/dl)
Change of biochemical metabolic parameters | Baseline and 4 weeks
  total proteins (g/dl)
Change of biochemical metabolic parameters | Baseline and 4 weeks
  transaminase alanine aminotransferase, aspartate aminotransferase (IU/L)
Change of biochemical metabolic parameters | Baseline and 4 weeks
  gamma glutamyl transferase, lipase and amylase (U/L)
Change of biochemical metabolic parameters | Baseline and 4 weeks
  Homocysteine (micromol/L)
Change of biochemical metabolic parameters | Baseline and 4 weeks
  Vitamin D and folic acid (ng/mL)
Change of biochemical metabolic parameters | Baseline and 4 weeks
  Vitamin B12 (pg/ml)
Change of inflammation markers | Baseline and 4 weeks
  C- Reactive protein (mg/dl)
Change of insulin resistance | Baseline and 4 weeks
  Homeostasis Model Assessment (HOMA) index
Change of satiating capacity | Every day for 4 weeks
  Haber score (point scale)
Change of anthropometric measures | Baseline and 4 weeks
  weight (kg)
Change of anthropometric measures | Baseline and 4 weeks
  Body mass index (Kg/m2)
Change of anthropometric measures | Baseline and 4 weeks
  calf circumference, waist circumference, arm circumference, hip circumference (cm)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda di Servizi alla Persona, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No